CLINICAL TRIAL: NCT06479980
Title: Pilot Study of Feasibility, Acceptability, Fit and Clinical Impact of a Single Session Narrative Psychotherapy Intervention to Reduce Wait Times in a Primary Care HIV Clinic
Brief Title: Single Session Narrative Therapy Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Akansha Vaswani Bye, Acting Assistant Professor, Department of Psychiatry and Behavioral Sciences, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00018612; 5P30MH123248-03 (NIH)
Record Dates: First submitted 2024-06-15; First posted 2024-06-28 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Mental Health Issue; HIV; Substance Use
Keywords: Brief narrative therapy; Implementation outcome; Stepped care; Psychotherapy; Integrated primary care
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Session Narrative Therapy Intervention (Experimental): A single 60-75 minute narrative therapy session with a trained licensed behavioral health provider will be offered to patients on the psychotherapy waitlist of an HIV primary care clinic.
  Interventions: Behavioral: Single Session Narrative Therapy

INTERVENTIONS:
Behavioral: Single Session Narrative Therapy — Single-session narrative psychotherapy intervention is an evidence-based strategy on a stepped care continuum that can assist patients in accessing care when they most need it and can lead to the most effective utilization of scarce resources. It offers a transdiagnostic, strengths, solution-oriented, and non-pathologizing intervention to address patients' behavioral health needs.
  Other Names: Brief Narrative Therapy

SUMMARY:
This pilot research study will provide timely access to behavioral health services through the provision of a single-session narrative therapy intervention. The goal of this 6-month study is to test the acceptability, feasibility, and fit of the intervention in an integrated primary care clinic serving people living with HIV.

DETAILED DESCRIPTION:
Single-session interventions are designed to address barriers to engaging in care and address the issues of long waitlists and limited provider availability. Offering a single session intervention soon after a referral is made is a strategy on a stepped-care continuum model that has been found to be an effective approach to manage population mental health needs. This study aims to 1) pre-pilot a single-session narrative therapy intervention with patients currently on the waitlist for psychotherapy services at an HIV primary care clinic to evaluate the acceptability of this treatment option for patients and the feasibility of proposed data collection followed by 2) a 6-month pilot study of the same intervention to evaluate intervention acceptability, fit, and impact on service and clinical outcomes. At the end of this study, patient and provider-level data on the utility of integrating a single-session psychotherapy service as part of the continuum of behavioral health services in an integrated care setting will be obtained, which the investigators can utilize to design a larger implementation-effectiveness trial.

ELIGIBILITY:
Patient Inclusion Criteria

* Adults (age 18 years and older) who are patients at [Blinded] Clinic
* Have agreed to participate in the single session intervention
* Ability to complete the interview and research surveys in English

Patient Exclusion Criteria:

* Participants with need for urgent mental health treatment (e.g., at imminent risk of suicide or harm to others; disabling symptom presentation)
* Inability to provide informed consent

Provider Inclusion Criteria:

* Adults (age 18 years and older)
* Referring providers at [Blinded] clinic (social worker, primary care physician, mental health professional etc.)
* Ability to complete the research survey or interview in English.

Provider Exclusion Criteria:

* Inability to provide informed consent
* Non-referring providers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | 0, 1 month
  The Patient Health Questionnaire-9 (PHQ-9) is a 9 item self-report measure used to screen for depression, diagnose it, monitor its severity, and measure treatment response. The PHQ-9 ranges from 0 to 27 points. A lower PHQ-9 total score indicates a better outcome.

SECONDARY OUTCOMES:
Generalized Anxiety Disorder- 7 (GAD-7) | 0, 1 month
  The Generalized Anxiety Disorder 7-item (GAD-7) is a brief self-report tool that measures anxiety symptoms based on the Diagnostic and Statistical Manual of Mental Disorders (DSM) criteria. The total score ranges from 0 to 21, with lower scores indicating better outcomes.
Remoralization Scale | 0,1 month
  The Remoralization Scale is a brief 12-item self-report tool that measures the level of morale. Score is a calculated mean that ranges from 1-4. Higher mean scores indicate a better outcome.
Social Connectedness Scale-Original (SCS-Original) | 0, 1 month
  The Social Connectedness Scale is an 8-item instrument which assesses the degree to which one feels connected to others in their social environment. Items are measured on a 6-point Likert scale (Strongly Agree-Strongly Disagree). Total scores range from 8 to 48 points. Higher total scores indicate a better outcome.
State-Trait Assessment of Resilience Scale (Trait sub-scale only) | 0, 1 month
  The State-Trait Assessment of Resilience Scale measures resilience using a state and trait approach, based on the conceptualization of resilience as being influenced by a combination of state and trait factors. This study will only measure the 'Trait' level of resilience, using the trait sub-scale (7-item instrument), which is construed as more distal and enduring. Total sum scores are calculated for the sub-scale and range from 7 to 28 points; higher scores indicate a better outcome.
Brief Services Evaluation | 0, 1 month
  The Brief Services Evaluation is a 6-item instrument which measures patients' assessment of their skills, ideas, and knowledge regarding the main problem/issue that brought them into counseling. Items are measured on a 6-point Likert scale (Strongly Disagree- Strongly Agree). Score is a calculated mean that ranges from 1-6. Higher mean scores indicate a better outcome.
Acceptability of Intervention Measure (AIM) | 1 month, Up to 8 months
  The Acceptability of Intervention Measure is a 4-item measure of perceived intervention acceptability. Items are measured on a 5-point Likert scale (Completely Disagree-Completely Agree). Score is a calculated mean that ranges from 1-5. Higher mean scores indicate a better outcome.
Intervention Appropriateness Measure (IAM) | Up to 8 months
  The Intervention Appropriateness Measure is a 4-item measure of perceived intervention appropriateness. Items are measured on a 5-point Likert scale (Completely Disagree-Completely Agree). Score is a calculated mean that ranges from 1-5. Higher mean scores indicate a better outcome.
Feasibility of Intervention Measure (FIM) | Up to 8 months
  The Feasibility of Intervention Measure is a 4-item instrument to assess perceived intervention feasibility. Items are measured on a 5-point Likert scale (Completely Disagree-Completely Agree). Score is a calculated mean that ranges from 1-5. Higher mean scores indicate a better outcome.

OTHER OUTCOMES:
Waitlist Evaluation Questionnaire | 0 months
  A 2-item questionnaire evaluating: a) if a patient would like to remain or be taken off the psychotherapy waitlist of [Blinded] clinic (yes or no) b) if the patient selects to remain on the waitlist, what service type they are seeking (Up to 3 single sessions scheduled when needed or 12-16 regularly scheduled sessions).
Modified Single Session Impressions and Feedback Tool- Adapted Version | 0 months
  The Single Session Impressions and Feedback tool is an 8-item post-session questionnaire which measures patient satisfaction and the degree to which the therapist adhered to key single session narrative therapy principles during the session. Items are measured a 7-point Likert scale (Strongly Disagree-Strongly Agree), where 7 represents the most positive score.
Single Session Consultation Feedback Form | 0 months
  The Single Session Consultation Feedback Form is a 5-item post-session questionnaire that measures patients' satisfaction with the therapy intervention. Items are measured on a Likert scale from 1 ("Not at all") to 5 ("Very much"), where 5 represents the most positive score.
Patient Participant Qualitative Interview | 1 month
  Qualitative interviews will be conducted with a subset of patient participants approximately 1 month after receiving the single session narrative therapy intervention. Interviews will be 30-45 minutes and address acceptability and appropriateness of the intervention; experiences being offered and participating in the intervention; facilitators and barriers to participating; what was particularly meaningful or useful about the intervention, and suggestions for improving the intervention.
Provider Participant Qualitative Interview | Up to 8 months
  Qualitative interviews will be conducted with a purposive sample of providers whose patients received the single session intervention to assess intervention acceptability, feasibility, and fit.

CONTACTS AND LOCATIONS:
Overall Officials: Akansha Vaswani-Bye, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Research subject's de-identified data will be shared through the National Institute of Mental Health Data Archive (NDA).
Time Frame: Data will made available in alignment with the first data submission date required by the National Institute of Mental Health Data Archive.
Access Criteria: Summary information on the data shared in NDA is available in the NDA Query Tool without the need for an NDA user account. To request access to record-level human subject data, a Data Access Request must be submitted.